CLINICAL TRIAL: NCT04434287
Title: Study of Prognostic Factors in Patients Admitted to ICU for Stroke
Acronym: REAVC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: REAVC ( 29BRC20.0062)
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Critically Ill
MeSH Terms: conditions — Stroke; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Outcome of stroke patients admitted to the intensive care unit the intensive care unit (ICU) is poor and haemorrhagic stroke, fixed dilated pupil(s) and GCS <10 are associated with increased mortality and poor functional outcome. However little is known about the impact of clinical events occuring during the ICU stay (ventilator acquired pneumoniae, shock, dysglycemia....).

The objective of this study was to determine the mortality rate and the functional outcomes of stroke patients admitted to ICU and to identify predictors of poor outcome in this population.

ELIGIBILITY:
Inclusion Criteria:

* acute stroke
* ICU admission for acute stroke
* 1 organ dysfunction : coma, shock, respiratory failure

Exclusion Criteria:

* refuse participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute stroke admitted to ICU in the Brest Teaching Hospital (Cavale Blanche) BREST (The Brest REgistry of STroke)
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Mortality | through ICU hospitalization, an average of one month

SECONDARY OUTCOMES:
Mortality | At 90 days
  Mortality
Functional outcome: Modified Rankin Score | at hospitalization discharge, an average of three months
  Modified Rankin Score (0: no symptoms at all; 6: dead)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two year and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.